CLINICAL TRIAL: NCT02421549
Title: Remote Interrogation of Implantable Cardiac Devices in Rural Emergency Departments
Brief Title: Remote Interrogation in Rural Emergency Departments
Acronym: REM RED
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 60054491
Record Dates: First submitted 2015-04-13; First posted 2015-04-20 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Disease; Cardiovascular Disease; Heart Failure; Arrhythmias, Cardiac
Keywords: Remote Monitoring; Remote Care; Cardiac Resynchronization Therapy; Pacemaker; Implantable Cardioverter Defibrillator
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interrogation with unpaired remote monitoring transmitter (Active Comparator): Interrogation with unpaired remote monitoring transmitter Interrogation with an unpaired remote monitoring transmitter for devices that are compatible.
  Interventions: Device: Unpaired remote monitoring transmitter
- Interrogation with Programmer (No Intervention): Interrogation with programmer Interrogation with programmer according to usual standard of care

INTERVENTIONS:
Device: Unpaired remote monitoring transmitter
  Other Names: SJM Merlin@home remote monitoring transmitter
  Arms: Interrogation with unpaired remote monitoring transmitter

SUMMARY:
A retrospective, multi-center, proof-of-concept study to evaluate the use of remote monitoring in rural emergency departments to decrease time to treatment decision for pacemaker and defibrillator patients using the St Jude Medical Merlin@home transmitter. The purpose of the study is to determine if utilization of remote monitoring technology in a rural emergency department may improve patient care.

Up to 10 rural ED sites will enroll a total of 200 patients. One hundred patients will be in the remote monitoring group comprised of patients with SJM devices compatible with the unpaired transmitter and 100 patients will be in the usual medical care group comprised of patients with SJM devices that are not compatible with the unpaired transmitter or that have a competitor's device.

ELIGIBILITY:
Inclusion Criteria:

1. Presents to Emergency Department with an implanted pacemaker or defibrillator.
2. Are 18 years of age or older.
3. Are willing and able to provide informed consent for study participation.
4. Are willing and able to complete a 30-60 day follow up phone call.

Exclusion Criteria:

1. Are unwilling to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Time to Clinical Specialist Treatment Decision | 1 day
  ED check in time to time of clinical specialist treatment decision.

SECONDARY OUTCOMES:
Health Care Utilization Rate | Within 30 days of initial ED visit
  Device related hospitalizations, ED visits and unscheduled office visits/urgent care visits within 30 days of the initial ED visit.

OTHER OUTCOMES:
Time to Device Interrogation | 1 day
  ED check in time until time of device interrogation

CONTACTS AND LOCATIONS:
Overall Officials: Ross Downey, MD, Principal Investigator — New Mexico Heart Institute, PA
Locations (1):
- New Mexico Heart Institute, Albuquerque, New Mexico, United States